CLINICAL TRIAL: NCT04561960
Title: Efficacy of Miswak When Compared to Fluoridated Toothpaste for the Maintenance of Oral Hygiene in Young Adults
Brief Title: Efficacy of Miswak in Oral Hygiene Maintenance
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Riyadh Elm University (Other)
Responsible Party: Principal Investigator, Sarah Samer Aburaisi, Principal Investigator, Riyadh Elm University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: FRP/2020/264
Record Dates: First submitted 2020-09-16; First posted 2020-09-24 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Dental Plaque
Keywords: miswak; siwak; S. persica; chew stick
MeSH Terms: conditions — Dental Plaque

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Active Comparator): Participants will be trained to perform oral hygiene using the modified bass technique.
  The participants will be asked to brush their teeth twice daily using a manual tooth brush and fluoridated toothpaste containing 1450ppm of fluoride
  Interventions: Drug: Fluoride toothpaste; Device: Toothbrush
- Miswak (Experimental): Participants will be trained to chew and condition a miswak stick Participants will be asked to use the miswak stick twice daily
  Interventions: Device: Miswak Stick
- Miswak Paste (Experimental): Participants will be trained to perform oral hygiene using the modified bass technique.
  The participants will be asked to brush their teeth twice daily using a manual tooth brush a non-fluoridated toothpaste containing miswak extract
  Interventions: Drug: Toothpaste Product; Device: Toothbrush

INTERVENTIONS:
Drug: Fluoride toothpaste — Fluoridated paste containing 1450ppm NaF
  Arms: Control
Drug: Toothpaste Product — Non Fluoridated toothpaste with extract of miswak ( Dabur, miswak tooth paste)
  Arms: Miswak Paste
Device: Toothbrush — Colgate classic clean Soft bristled toothbrushes, 19.05 x 1.27 x 1.91 cm
  Arms: Control; Miswak Paste
Device: Miswak Stick — A miswak stick of 15 cm length
  Arms: Miswak

SUMMARY:
Miswak has been recommended by world health organization for oral hygiene because of its availability, beneficial effect and affordability. The popularity of Miswak in Arab countries has meant that there have been several studies that have confirmed the ability of miswak to provide effective mechanical and chemical cleansing when used as an adjunct to other oral hygiene aids.

Fluoridated tooth paste and manual tooth brushes have been the standard of clinical preventive dental care for over 50 years.However, the objection to the use of fluorides by some parents has meant that these pastes are not universally accepted.

There are several non-fluoridated pastes available in the market that include the extract of miswak. There are few studies that have compared these pastes to fluoridated pastes and to miswak as a stand alone agents.

Miswak has been recommended by world health organization in 1987 for oral hygiene because of its availability, beneficial effect and affordability.

It has been stated that "Several clinical studies have confirmed that the mechanical and chemical cleansing efficiency of miswak chewing sticks are equal and at times greater than that of the toothbrush" this was mentioned and reviewed that it is in fact right but only when used in a regular constant matter with a proper and effective way of plaque removal. This study aims to use a cross over model to study the effectiveness of miswak as a stand alone agent in maintaining oral hygiene in young adults and compare it miswak containing toothpastes and fluoridated toothpastes when used with a manual tooth brush.

DETAILED DESCRIPTION:
Oral hygiene is the key of maintaining human's mouth at a state of equilibrium and free of diseases (e.g. cavities, dental decay, gingivitis, halitosis). Poor oral hygiene can significantly affect the quality of life and has a considerable influence on diet, sleeping, social communication, psychological status, and by being less productive at work.

Therefore, oral hygiene is essential for general health and well-being. Oral hygiene measures include toothbrush which is the most commonly used method for plaque control. However, miswak is a commonly used method in many developing countries.

Miswak has a widespread among religious, rural and developing countries for its spiritual impact since the use of miswak was advised by prophet mohammed (peace be upon him) centuries ago as he said "had I not thought it difficult for my ummah, I would have commanded them to use miswak before every prayer".

Miswak has been recommended by world health organization for oral hygiene because of its availability, beneficial effect and affordability. Previous chemical examinations changed our idea in Miswak which showed us that miswak sticks contain natural ingredients which benefits our oral health. Miswak extracts appear to have different beneficial biological properties like anti-bacterial and anti-fungal effects which will play a high role in oral hygiene measures.

Multiple researches suggested that miswak has anti-cariogenic effects. several studies concluded that Chewing sticks (miswak) has revealed parallel and at times greater mechanical and chemical cleansing of oral tissues as compared to a toothbrush.

The popularity of Miswak in Arab countries has meant that there have been several studies that have confirmed the ability of miswak to provide effective mechanical and chemical cleansing when used as an adjunct to other oral hygiene aids. In a previous study found that the periodontal health of miswak users was better than the periodontal health of manual toothbrush users, also it was concluded that miswak is more effective than tooth brushing for reducing plaque and gingivitis when preceded by professional instruction regarding its correct application.

Another research reported the opposite thing, Punit Patel and S. Shruthi studied the clinical effects of miswak as an adjunct to tooth brushing on gingivitis clearly and they find that the indication of miswak cannot replace the toothbrush, but can be used an adjunct to toothbrush, utilizing the mechanical efficacy of toothbrush and chemical effects of miswak.

However, it was concluded that "The use of S. persica miswak alone or in combination with conventional toothbrushes, when performed judiciously, will result in superior oral health and hygiene." Fluoridated tooth paste and manual tooth brushes have been the standard of clinical preventive dental care for over 50 years. However, the objection to the use of fluorides by some parents has meant that these pastes are not universally accepted.

There is a lot of controversy whether the miswak alone can be used for effective plaque removal and good gingival health or should it be only used as an adjunct to tooth brushing.

In this study we will determine whether the miswak can be used as the chief tool in oral health rather than an adjunct to tooth brushing. We will also determine whether toothpaste using the miswak extract can be as effective as the normal fluoridated toothpaste.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults
* Able to perform their own oral hygiene
* Dental students

Exclusion Criteria:

* Active Dental Caries
* Uncontrolled chronic medical conditions
* History of drug and/or treatment that reduces salivary flow
* Currently undergoing orthodontic treatment
* Missing index teeth #16, #12, #24, #36, #32, #44

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Base line Plaque Score | Baseline
  Silness-Löe Index: #16, #12, #24, #36, #32, #44Missing teeth are not substituted. 0-3, 0 being absent from plaque
Plaque Score change at 1 week | One week
  Silness-Löe Index: #16, #12, #24, #36, #32, #44Missing teeth are not substituted. 0-3, 0 being absent from plaque
Plaque Score change at 2 weeks | Two weeks
  Silness-Löe Index: #16, #12, #24, #36, #32, #44Missing teeth are not substituted. 0-3, 0 being absent from plaque
Baseline Bleeding Score | Baseline
  Gingival Index (Loe & Silness 1963): #16, #12, #24, #36, #32, #44Missing teeth are not substituted. 0-4 . 0 being absent from inflammation
Bleeding Score change at 1 week | One week
  Gingival Index (Loe & Silness 1963): #16, #12, #24, #36, #32, #44Missing teeth are not substituted. 0-4 . 0 being absent from inflammation
Bleeding Score change at 2 weeks | Two weeks
  Gingival Index (Loe & Silness 1963): #16, #12, #24, #36, #32, #44Missing teeth are not substituted. 0-4 . 0 being absent from inflammation

SECONDARY OUTCOMES:
Presence of White spot lesions | Two weeks
  Visual Initial signs of dental caries

CONTACTS AND LOCATIONS:
Overall Officials: Omar Alkadhi, MSc, Study Chair — Head of IRB, REU; Sarah S Aburaisi, MSc, Principal Investigator — Assistant Professor, prothetic dental department, REU
Locations (1):
- Riyadh Elm University, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hawkins BF, Kohout FJ, Lainson PA, Heckert A. Duration of toothbrushing for effective plaque control. Quintessence Int. 1986 Jun;17(6):361-5. No abstract available. PMID 3460112
- [Result] Elvin-Lewis M. The therapeutic potential of plants used in dental folk medicine. Odontostomatol Trop. 1982 Sep;5(3):107-17. No abstract available. PMID 6962424
- [Result] Patel PV, Shruthi S, Kumar S. Clinical effect of miswak as an adjunct to tooth brushing on gingivitis. J Indian Soc Periodontol. 2012 Jan;16(1):84-8. doi: 10.4103/0972-124X.94611. PMID 22628969
- [Result] Al-Otaibi M, Al-Harthy M, Gustafsson A, Johansson A, Claesson R, Angmar-Mansson B. Subgingival plaque microbiota in Saudi Arabians after use of miswak chewing stick and toothbrush. J Clin Periodontol. 2004 Dec;31(12):1048-53. doi: 10.1111/j.1600-051X.2004.00618.x. PMID 15560804
- [Result] Halawany HS. A review on miswak (Salvadora persica) and its effect on various aspects of oral health. Saudi Dent J. 2012 Apr;24(2):63-9. doi: 10.1016/j.sdentj.2011.12.004. Epub 2012 Jan 28. PMID 23960531
- [Result] Haque MM, Alsareii SA. A review of the therapeutic effects of using miswak (Salvadora Persica) on oral health. Saudi Med J. 2015 May;36(5):530-43. doi: 10.15537/smj.2015.5.10785. PMID 25935172
- [Result] Devi, Aruna M.; Hampannavar, Pooja; Radha, G.; Kadanakuppe, Sushi; Nagashree, S. R.; Kumar, Vinod A. (2011) Comparing the Efficacy of Plaque Removal between Salvadora persica (Miswak) and Manual Toothbrush in 12 to 15 Years School Children. World Journal of Dentistry, 2(1), pp. 29-33.
- [Result] Norton MR, Addy M. Chewing sticks versus toothbrushes in West Africa. A pilot study. Clin Prev Dent. 1989 May-Jun;11(3):11-3. PMID 2605858
- [Result] Malik AS, Shaukat MS, Qureshi AA, Abdur R. Comparative effectiveness of chewing stick and toothbrush: a randomized clinical trial. N Am J Med Sci. 2014 Jul;6(7):333-7. doi: 10.4103/1947-2714.136916. PMID 25077082
- [Result] World Health Organization. (1997). Oral health surveys: basic methods, 4th ed. World Health Organization
- [Result] Darout IA, Skaug N, Albandar JM. Subgingival microbiota levels and their associations with periodontal status at the sampled sites in an adult Sudanese population using miswak or toothbrush regularly. Acta Odontol Scand. 2003 Apr;61(2):115-22. doi: 10.1080/00016350310002784. PMID 12790510